CLINICAL TRIAL: NCT03469115
Title: New Insights Into the Metabolic Syndrome: the Role of Alpha Defensin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HYMC-15-18
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Adolescents aged 13-17 will be divided into two groups according to BMI (body mass index)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI above 95% (Active Comparator): Serum blood will be taken from obese youths with suspected metabolic syndrome
  Interventions: Diagnostic Test: Serum blood
- BMI below 3% (Active Comparator): Serum blood will be taken from slim youths
  Interventions: Diagnostic Test: Serum blood

INTERVENTIONS:
Diagnostic Test: Serum blood — Serum blood test for laboratory analysis to determine level of alpha defensin

SUMMARY:
The purpose of this study is to find out if there is a connection between a higher level of peptide alpha defensin in blood serum with the metabolic profile of adolescents aged 13-17.

ELIGIBILITY:
Inclusion Criteria:

* Youths with metabolic syndrome (BMI above 95%)
* Youths with BMI below 3%

Exclusion Criteria:

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Alpha defensin level | 2 hours
  Alpha defensin level above 12ng/microliter

CONTACTS AND LOCATIONS:
Overall Officials: Eias Kassem, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No